CLINICAL TRIAL: NCT03104309
Title: Can the Effect of Levonorgestrel Intrauterine System for Treatment of Adenomyosis be Predicted at Baseline Visit?
Brief Title: Levonorgestrel Intrauterine System and Adenomyosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mohammed Khairy Ali, Dr, Assiut University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LNG_ADENO
Record Dates: First submitted 2017-04-03; First posted 2017-04-07 (Actual); Last update posted 2017-04-14 (Actual); Status verified 2017-04

CONDITIONS: Adenomyosis
MeSH Terms: conditions — Adenomyosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Levonorgestrel intrauterine system (Other)
  Interventions: Device: Levonorgestrel intrauterine system

INTERVENTIONS:
Device: Levonorgestrel intrauterine system — Levonorgestrel intrauterine system for adenomyosis

SUMMARY:
Adenomyosis is defined when the endometrial tissue (gland and stroma) is present within the myometrium . The depth of endometrial penetration which uses in diagnosis of adenomyosis not yet agreed; opinions range from one high power field to 25% of the myometrial thickness. It is a common condition in women aged 40-50 years and is considered an important cause of dysmenorrhea and menorrhagia in around 65 % of cases.

Until past few years; hysterectomy was the suggested definitive treatment, however; this may not be acceptable to women not willing to loss their fertility. Many treatment lines were studied and proved their beneficial effect on adenomyosis such as GnRH agonists, danazol, combined oral contraceptive pills, dienogest and finally endometrial ablation. However, these line of treatment are not commonly used because high incidence of side effects and relatively high cost of some of them.

The levonorgestrel-releasing intrauterine system (LNG-IUS) was emerged as an effective line for treatment of adenomyosis associated pain and bleeding. It can successfully, within 6 to 12 months, down-regulate the estrogen receptors in adenomyotic tissues which lead to decidualization and atrophy of the adenomyosis .

In fact, some adenomyotic women respond well to LNG-IUDs and show high acceptability and satisfaction, on the other hand; a group of women may not respond to LNG-IUDs and opt to remove it and start a new medical or surgical option for treatment.

However, factors related to LNG-IUS effectiveness in patients with adenomyosis were not well available. Only one report states that a large uterine volume could be a factor associated with LNG-IUS treatment discontinuation in adenomyotic patient.

For this reason; the prediction of the responsiveness to LNG-IUS is interesting issue which should be addressed. The present study examines the hypothesis that patient's data reported at baseline visit before using LNG-IUSfor controlling pain/bleeding with adenomyosis can help the prediction of the responsiveness for this important line of treatment at 6 months follow up visit. Up to our knowledge; no clinical trial had been registered or conducted to predict the responsiveness for LNG-IUS in controlling the pain/ bleeding with adenomyosis.

ELIGIBILITY:
Inclusion Criteria:

* adenomyosis
* request for contraception
* resident in the nearby vicinity to make the follow-up easy and feasible

Exclusion Criteria:

* history of ectopic pregnancy
* puerperal sepsis
* pelvic inflammatory disease
* evidence of coagulopathy
* abnormalities of the uterine cavity

Ages: 20 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2015-06 (Actual); Primary Completion 2016-07 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
number of bleeding days per months | 6 months
The degree of pain perception by visual analogue scale | 6months

IPD SHARING:
Plan to Share IPD: Yes